CLINICAL TRIAL: NCT00093223
Title: A Phase II Safety Study of Systemic Nanoparticle Paclitaxel (ABI-007)for In-Stent Restenosis
Brief Title: A Safety Study of ABI-007 for In-Stent Restenosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVR001
Record Dates: First submitted 2004-10-04; First posted 2004-10-07 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Angina Pectoris; Coronary Artery Disease
Keywords: In-Stent Restenosis
MeSH Terms: conditions — Angina Pectoris; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 35mg/m^2 infusion time is 3.5 minutes
  Interventions: Drug: Paclitaxel Nanoparticle Albumin Bound
- 2 (Experimental): 2 doses of 35mg.m^2 with the second dose given 2 months later
  Interventions: Drug: Paclitaxel Nanoparticle Albumin Bound

INTERVENTIONS:
Drug: Paclitaxel Nanoparticle Albumin Bound — Single or duel doses of 35mg/m^2 ABI-007, administered IV, administered after placement of denovo stent(s).
Drug: Paclitaxel Nanoparticle Albumin Bound
  Arms: 1
Drug: Paclitaxel Nanoparticle Albumin Bound — 35mg/35 infusion time is 3.5 minutes
  Arms: 2

SUMMARY:
This trial will treat patients with a new chemotherapeutic medicine who have undergone a successful and uncomplicated de novo stent placement in up to two native coronary arteries. The purpose of the trial is to determine the appropriate dose of the new medicine for future trials and to evaluate the incidence of treatment-emergent adverse events and serious adverse events.

DETAILED DESCRIPTION:
See inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Undergone a successful and uncomplicated de novo stent placement in up to two native coronary arteries
* Diagnosis of angina pectoris
* At least 18 yrs old
* If female, negative pregnancy test, non-lactating, and agree to utilize methods to prevent pregnancy
* No previous treatment for In-Stent Restenosis
* Patient agrees to comply with follow-up evaluation
* Informed Consent obtained
* Target vessel at least 3 mm diameter
* Total stent less than 25 mm
* Left ventricular ejection fraction at least 30%
* No more than a single stent will be used per lesion
* No more than one stented lesion per vessel with the exception that 2 lesions in a single vessel are allowable if covered by less than 25 mm of continuous stent
* By Intravascular Ultrasound (IVUS), stent is fully opposed and has a minimum diameter of 3 mm or an in-stent luminal area of at least 7 mm2
* TIMI 3 coronary flow post-stenting
* No angiographic evidence of thrombus post-stenting

General Exclusion Criteria:

* More than two lesions treated with Percutaneous Coronary Intervention (PCI) or it is anticipated that additional lesions will require treatment within two months
* Previous PCI within preceding three months
* Previous participation in another study within 30 days
* Life expectancy less than 12 months
* Factors making follow-up difficult
* Intended surgical intervention within 6 months of study participation
* Investigator decision that patient is unsuitable
* Recipient of heart transplant
* Q wave or non-Q wave Myocardial Infarction (MI) with documented total CK greater than 2X normal upper limits within the preceding 24 hrs and the CK and CK-MB enzymes remain above normal at the time of the procedure
* Cardiogenic shock
* May refuse blood transfusion
* Gastro-intestinal bleeding within past 3 months
* Platelet count less than 100,000 cells/mm3
* Impaired renal function
* Known allergies/hypersensitivity to aspirin, clopidogrel bisulfate, and/or stainless steel

Exclusion Criteria Related to Angioplasty:

* Intervention for another lesion occurred within 90 days or is planned for within 60 days after the index procedure
* Stent is located in a coronary bypass
* Unprotected left main disease with greater than 50% stenosis
* Lost a side branch greater than 2 mm during stenting procedure
* Angiographic evidence of thrombus post-stenting
* Prior stent within 5 mm of target lesion
* Left ventricular ejection fraction less than 30%
* Greater than 50% stenosis proximal or distal to target lesion
* Malposition, dissection, or unmasking of a significant narrowing in the inflow or outflow area of the implanted stent
* Patient has received a drug coated stent as part of this procedure

Exclusion Criteria Related to ABI-007:

* Absolute neutrophil count is less than 1500 cells/mm3
* Platelet count is less than 100,000 cells/mm3
* Bilirubin greater than 1.5 mg/dl or SGOT and SGPT greater than 2.5X upper limit of normal or alkaline phosphatase greater than 2.5X upper limit of normal
* Creatinine greater than 2.5X upper limit normal
* Pre-existing peripheral neuropathy of NCI toxicity Criteria Scale of Grade greater than 1
* Immunosuppressed or has HIV or AIDS
* Hypersensitivity to Taxane

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2001-09-01 (Actual); Primary Completion 2007-12-01 (Actual); Study Completion 2007-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events and serious adverse events. | 6 months
Major Adverse Cardiac Events at 2 months following the stent procedure. | 2 months
Safety and tolerability for ABI-007 | 2 Years

SECONDARY OUTCOMES:
Evaluation of restenosis at 6 months. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: José Iglesias, MD, Study Director — Celgene Corporation
Locations (1):
- Abraxis BioScience, Inc., Durham, North Carolina, United States